CLINICAL TRIAL: NCT05927428
Title: An Open-Label, Multi-Center, Phase 2 Dose Ranging Study of BRM424 Ophthalmic Solution in Patients With Neurotrophic Keratitis (NK)
Brief Title: Assessment of the Initial Efficacy and Safety of BRM424 Ophthalmic Solutions in Patients With Neurotrophic Keratitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BRIM Biotechnology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRM424-21-C001
Record Dates: First submitted 2023-05-31; First posted 2023-07-03 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Neurotrophic Keratitis

STUDY DESIGN:
Intervention Model Description: Open-label, Randomized Study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BRM424 Ophthalmic Solution - Dose1 (Active Comparator)
  Interventions: Drug: BRM424 Ophthalmic Solution - Dose1
- BRM424 Ophthalmic Solution - Dose2 (Active Comparator)
  Interventions: Drug: BRM424 Ophthalmic Solution - Dose2

INTERVENTIONS:
Drug: BRM424 Ophthalmic Solution - Dose1 — A topical drop of BRM424 ophthalmic solution.
  Arms: BRM424 Ophthalmic Solution - Dose1
Drug: BRM424 Ophthalmic Solution - Dose2 — A topical drop of BRM424 ophthalmic solution.
  Arms: BRM424 Ophthalmic Solution - Dose2

SUMMARY:
The objective of this study is to obtain initial efficacy of BRM424 in patients with Stage 2 and Stage 3 NK and evaluate safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Patients with NK Stage 2 (PED) or Stage 3 (corneal ulcer);

Exclusion Criteria:

* Any active ocular infection (bacterial, viral, fungal or protozoal) or active ocular inflammation not related to NK;
* Anticipated need to use therapeutic contact lenses or contact lens wear for refractive correction during the 28-days Treatment Period in the eye(s) with NK;
* Be a woman of childbearing potential who is not using an acceptable means of birth control;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving complete healing of the PED or corneal ulcer determined by corneal fluorescein staining | at or before 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmington Eye, Leland, North Carolina, United States